CLINICAL TRIAL: NCT06075290
Title: Application of Two Different Follow-up Methods for Neonatal Jaundice in the Prevention of Severe Hyperbilirubinemia
Brief Title: the Difference of Follow-up Methods of Neonatal Jaundice
Acronym: NJFU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEO20230802
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Neonatal Jaundice
Keywords: neonatal jaundice; follow-up; internet plus model; severe hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia | interventions — Models, Biological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: Intelligent jaundice instrument and Internet plus system for home monitoring and remote follow-up
  Interventions: Behavioral: internet plus model
- control group: follow-up by conventional methods ； hospital or community follow-up depending on arrangement
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: internet plus model — Intelligent transcutaneous bilirubin meter and Internet plus model for neonatal jaundice monitoring at home and remote follow-up
  Groups: Observation group
Behavioral: control — follow-up by conventional methods; hospital or community follow-up depending on arrangement
  Groups: control group

SUMMARY:
The goal of this observational study is to compare the effectiveness and efficiency for precaution of severe hyperbilirubinemia in neonate by different follow-up methods of neonatal jaundice. There are two kinds of follow-up methods in the investigators clinical practice. The one is internet plus follow-up model, the other is conventional clinic follow-up method. Parents of the participant neonates can choose one by themselves. After parents of the participant signed informed consent, the investigators recorded several information including severe hyperbilirubinemia, length of phototherapy, follow-up times, et al. Then the investigators analysed these data in order to know what kind of follow-up method is better to prevent severe hyperbilirubinemia and more easy to be accepted.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≥ 28 weeks, corrected gestational age ≤ 44 weeks;
2. Presence of skin yellowing, percutaneous measurement of jaundice or serum bilirubin concentration less than the phototherapy warning value for the same gestational age and day age group;
3. The vital signs are stable and meet the discharge requirements;
4. Agree to participate in this project and sign an informed consent form;
5. Parents have a certain understanding ability to cooperate in this study;

Exclusion Criteria:

1. Direct bilirubin ≥34mmol/L;
2. Increased hepatic enzyme level more than twice of normal value;
3. Those infants who have developed bilirubin encephalopathy or neurological damage due to other reasons before follow-up;
4. Unable to continue follow-up due to other diseases.

Ages: 0 Days to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neoborns, gestational age ≥ 28 weeks, corrected gestational age ≤ 44 weeks
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe hyperbilirubinemia | 10,01,2023 to 10,01,2024
  The peak concentration of serum bilirubin is more than the exchange criteria of same gestational age and day age group
Newborn follow-up rate | 10,01,2023 to 10,01,2024
  Number of newborns who completed the follow-up program/total number of follow-up newborns

SECONDARY OUTCOMES:
Incidence rate of acute bilirubin encephalopathy | 10,01,2023 to 10,01,2024
  Number of infants with acute bilirubin encephalopathy/total number of follow-up newborns
Mean bilirubin level at admission | 10,01,2023 to 10,01,2024
  sum total serum bilirubin of hospitalized newborns at admission/Total number of hospitalized newborns
Follow-up satisfaction | 10,01,2023 to 10,01,2024
  Parents' comments of participating in the study
Average economic cost of treatment | 10,01,2023 to 10,01,2024
  Treatment and transportation costs and so on

CONTACTS AND LOCATIONS:
Overall Officials: Rong Chen, doctor, Principal Investigator — Guizhou Provincial People's Hospital
Locations (3):
- China (3):
  - People's Hospital of Anshun City Guizhou Province, Anshun, Guizhou
  - The First Affiliated Hospital of Guizhou University of Chinese, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou

IPD SHARING:
Plan to Share IPD: Yes
Scientific publishing
Supporting Information: Study Protocol, CSR
Time Frame: 12,31,2025
Access Criteria: open